CLINICAL TRIAL: NCT06387420
Title: A Phase 1b/2 Study of AK117 (Anti-CD47 Antibody) in Combination With Azactidine Plus Venetoclax in Patients With Acute Myeloid Leukemia
Brief Title: A Study of AK117 in Combination With Azactidine Plus Venetoclax in Patients With Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK117-206
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: ACUTE MYELOID LEUKEMIA; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK117+Azacitidine+Venetoclax (Experimental): Phase Ib: Subjects will receive: A117: different doses on every 2 weeks, azacitidine: 75 mg/m^2 on Days 1-7 each cycle, venetoclax: 100 mg on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, 400 mg on Cycle 1 Day 3 and daily thereafter;
  Phase II: Subjects will receive: AK117: the recommended Phase 2 dose (RP2D) on every two weeks, azacitidine: 75 mg/m^2 on Days 1-7 each cycle, venetoclax: 100 mg on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, 400 mg on Cycle 1 Day 3 and daily thereafter.
  Interventions: Drug: AK117; Drug: Azacitidine; Drug: Venetoclax
- Placebo+Azacitidine+Venetoclax (Placebo Comparator): Phase II: Subjects will receive: placebo: the recommended Phase 2 dose (RP2D) on every two weeks, azacitidine: 75 mg/m^2 on Days 1-7 each cycle, venetoclax: 100 mg on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, 400 mg on Cycle 1 Day 3 and daily thereafter.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Other: Placebo

INTERVENTIONS:
Drug: AK117 — Subjects receive AK117 intravenously.
  Arms: AK117+Azacitidine+Venetoclax
Drug: Azacitidine — Subjects receive azacitidine subcutaneously.
Drug: Venetoclax — Subjects receive venetoclax orally.
Other: Placebo — Subjects receive placebo intravenously.
  Arms: Placebo+Azacitidine+Venetoclax

SUMMARY:
This is a phase 1b/2 study. All patients are diagnosed with Acute Myeloid Leukemia (AML), Eastern Cooperative Oncology Group (ECOG) performance status 0-3. The purpose of this study is to evaluate the safety and efficacy of AK117 + azacitidine + venetoclax in subjects with AML.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at the time of enrolment.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0~3, and 0~2 are required for subjects ≥75 years old.
* Has a life expectancy of at least 12 weeks.
* Diagnosed as AML diagnosed according to WHO 2022 criteria.
* Has adequate organ function.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Diagnosed with acute promyelocytic leukemia, BCR-ABL1-positive AML, myeloid sarcoma, mixed phenotype acute leukemia (MPAL), accelerated phase or blast crisis of Chronic Myeloid Leukemia.
* has central nervous system leukemia (CNSL).
* Favorable risk cytogenetics such as t(8;21), inv(16) or t(16;16) or t(15;17) as per the National Comprehensive Cancer Network (NCCN) Guidelines Version 6, 2023 for AML.
* Previously diagnosed with another malignancy or have any evidence of residual disease.
* Previous allogeneic hematopoietic stem cell transplant (allo-HSCT).
* Prior treatment with any B-cell lymphoma 2 (Bcl-2) inhibitors, anti-CD47 or anti-SIRPα (signal regulatory protein alpha) agent.
* Use strong or moderate cytochrome P450 (CYP) 3A inducers systemically within one week prior to enrollment, or currently require long-term treatment with a moderate to strong CYP3A inducer.
* Previously diagnosed with MDS and treated with demethylating drugs.
* Patients with known cardiopulmonary disease defined as unstable angina, clinically significant arrhythmia, congestive heart failure (New York Heart Association Class III or IV), decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders.
* Other conditions where the investigator considers the patient inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-04-29 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of participants with dose limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  Any untoward medical occurrence in a subject within the first cycle, considered related to the study treatment
Phase 1b/2: Number of participants with adverse events (AEs) | Up to approximately 2 years.
  Any untoward medical occurrence in a subject, temporally associated with the use of study treatment, whether or not considered related to the study treatment
Phase 1b/2: Composite complete remission rate (CCR) | Time Frame: Up to approximately 2 years
  The proportion of subjects achieving complete remission (CR) , complete remission with partial hematologic recovery (CRh) or complete remission with incomplete hematologic recovery (CRi) per European LeukemiaNet (ELN) 2022 criteria

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 2 years
  The proportion of subjects with recorded response per European LeukemiaNet (ELN) 2022
Time to response (TTR) | Up to approximately 2 years
  Time from cycle 1 day 1(C1D1) to the first recorded response
Time to CCR (TTCCR) | Up to approximately 2 years
  Time from C1D1 to the first recorded CR, CRh or CRi
Duration of response (DoR) | Up to approximately 2 years
  Time from the first recorded response until disease progression, relapse, or death due to any cause, whichever occurs first
Duration of CCR (DoCCR) | Up to approximately 2 years
  Time from the first recorded CR, CRh or CRi until disease progression, relapse, or death due to any cause, whichever occurs first
Rate of CCR Without Minimal Residual Disease (CCR MRD-) | Up to approximately 2 years
  The proportion of subjects achieving CR, CRh or CRi with MRD-negative status per ELN 2022 criteria.
Event-free survival (EFS) | Up to approximately 2 years
  Time from C1D1 until disease progression, relapse, or death due to any cause, whichever occurs first
Overall survival (OS) | The time from C1D1 until death due to any cause
  Up to approximately 2 years
Peak of Serum Concentration (Cmax) | Up to approximately 2 years
  Maximal serum concentrations of AK117 in individual subjects at different time points after AK117 administration
Anti-drug antibody (ADA) | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies
Receptor occupancy (RO) | Up to approximately 2 years
  CD47 occupancy rate on peripheral blood T cells and red blood cells before and after AK117 administration

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, China

IPD SHARING:
Plan to Share IPD: No